CLINICAL TRIAL: NCT01940926
Title: Diagnostic Performance and Evaluation Efficacy of 68Ga-BNOTA-PRGD2 PET/CT in Patients With Rheumatoid Arthritis
Brief Title: 68Ga-BNOTA-PRGD2 PET/CT in Patients With Rheumatoid Arthritis
Acronym: GRGDRA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM07
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; angiogenesis; 68Ga-PRGD2; 18F-FDG; positron emission tomography/computed tomography
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 68gallium-BNOTA-PRGD2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-BNOTA-PRGD2 (Experimental): In patients with RA, single dose intravenous injection of nearly 111 MBq 68Ga-BNOTA-PRGD2 will be given at 30 minutes before PET/CT scanning to determine 68Ga-BNOTA-PRGD2 uptake in joints.
  Interventions: Drug: 68Ga-BNOTA-PRGD2

INTERVENTIONS:
Drug: 68Ga-BNOTA-PRGD2 — Single dose intravenous injection of nearly 111 MBq 68Ga-BNOTA-PRGD2 at 30 minutes before PET/CT scanning
  Other Names: 68Ga-p-SCN-Bn-NOTA-PEG3-RGD2

SUMMARY:
This is an open-label positron emission tomography/computed tomography ( PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-BNOTA-PRGD2 in rheumatoid arthritis (RA) patients. A single dose of nearly 111 MBq 68Ga-BNOTA-PRGD2 (≤ 40 µg BNOTA-PRGD2) will be intravenously injected into patients with RA. Visual and semiquantitative method will be used to assess the PET/CT images. Whole body 18F-FDG PET/CT will be performed for comparison.

DETAILED DESCRIPTION:
The Alpha(v)beta3 integrin, one of the most prominent members of integrin superfamily, is trans-membrane heterodimeric proteins which mediate cell-cell and cell-extracellular matrix adhesion. Integrin alpha(v)beta3 receptor plays an pivotal role in promoting, sustaining and regulating the angiogenesis and was identified as a marker of angiogenic vascular tissue. Cyclic arginine-glycine-aspartic acid (RGD) peptides was identified as a key integrin recognition motif which could strongly bind to integrin alpha(v)beta3 and inhibit new blood vessel formation. Animal study in antigen induced arthritis demonstrated that intra-articular administration of a cyclic RGD antagonist of alpha(v)beta3 leading to inhibition of cell infiltrate, synovial angiogenesis, pannus formation, cartilage erosions and even diminishing arthritis severity. For these properties, RGD peptide-based multimodality molecular probes have been developed for noninvasive imaging by targeting integrin alpha(v)beta3. And compared with 18F-FDG PET/CT, radiolabeled RGD imaging is a promising approach to visualize angiogenesis and provide a therapeutic target for anti-angiogenetic and anti-integrin therapy.

For the further interests in clinical translation of 68Ga-BNOTA-PRGD2, an open-label PET/CT study was designed to investigate the diagnostic performance and evaluation efficacy of 68Ga-BNOTA-PRGD2 in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilled the 1987 revised criteria of the American College of Rheumatology (ACR) for RA;
* Males and females, ≥18 years old

Exclusion Criteria:

* Concurrent medical conditions of other autoimmune diseases
* Latent or active joint infection or joint injury
* Renal dysfunction (serum level of creatinine more than 1.2 mg/dL)
* Females planning to bear a child recently or with childbearing potential
* Known severe allergy or hypersensitivity to intravenous radiographic contrast
* Inability to lie still for the entire imaging time because of cough, pain, etc
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Semiquantitative assessment (Standardized Uptake Values = SUVs) of lesion | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of 68Ga-BNOTA-PRGD2 will be measured using a volume-of-interest method.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 1 year
  Adverse events within 5 days after intravenous injection of 68Ga-BNOTA-PRGD2 and PET/CT scanning will be collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Z, Yin Y, Zheng K, Li F, Chen X, Zhang F, Zhang X. Evaluation of synovial angiogenesis in patients with rheumatoid arthritis using (6)(8)Ga-PRGD2 PET/CT: a prospective proof-of-concept cohort study. Ann Rheum Dis. 2014 Jun;73(6):1269-72. doi: 10.1136/annrheumdis-2013-204820. Epub 2014 Feb 14. PMID 24532680